CLINICAL TRIAL: NCT05848752
Title: On-line Crowdsourcing of Multi-Timescale Inference Strategies
Brief Title: Studies of Human Inference Using On-line Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Pennsylvania (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Tahra Eissa, Research Associate, University of Colorado, Boulder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-0065
Record Dates: First submitted 2023-04-19; First posted 2023-05-08 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior | interventions — Psychophysics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Environmental Feature Experiment (Experimental)
  Interventions: Behavioral: psychophysics

INTERVENTIONS:
Behavioral: psychophysics — Subjects will be shown a pair of jars each filled with the same absolute number but different ratios of red/blue balls. Three blocks of trials exist, short-term inference (subjects must identify which of the equally likely jars is currently in use), long-term inference (subjects must predict the subsequent jar in use on the next trial, where jar switches are correlated across trials), or multi-timescale inference (subjects must both report the current jar and predict the subsequent jar, combining the short and longterm inferences). Subjects will draw balls as many balls as they wish with replacement (free response) during the short-term and multi-timescale blocks but will know the current jar in use for long-term inference.

SUMMARY:
The investigators will record behavioral responses from human participants on crowdsourcing platform Prolific to identify the decision strategies humans apply short-term, long-term, and multi timescale (across both timescales) inference tasks. Participants will perform a Jar Switching Task (described in Research Strategy Aim 1- "Jar Switching Task") in which balls are drawn with replacement from one of two known jars. The current jar in use switches based on an underlying change rate across trials. Subjects must perform three task blocks: 1) report the current jar in use (short-term inference), 2) predict the subsequent jar (long-term inference), and 3) both report and predict the jars (multi-timescale inference). The investigators will record these responses, the number (and sequence) of balls drawn, and the response time (time from the end of trial until the response) for each trial. Subjects will perform all blocks (parameters and number of blocks to be determined by inference model development and testing prior to task development) so that we can compare responses at each timescale. Since participants participate voluntarily for small sums of money (around $10/ hour based on duration of task) and the investigators' previous studies have collected over 200 subjects in a matter of days, they will aim to record behavioral data from 1000 subjects. This number allows them to address the broad range of subject variability expected using Bayesian statistical methods such as Bayes factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult Prolific participants who have a 95% approval rating and achieve a minimum score of 80% on our pre-test,
* Speak fluent English
* Are in the US.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Binary Behavioral Decision Responses | Through task completion on each task trial, approximately 1-5x/ minute for approximate 30 minutes
  Subject- provided choices (responses on the computer) between two presented options

CONTACTS AND LOCATIONS:
Overall Officials: Tahra Eissa, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The task structure will be preregistered to Open Science Framework (OSF) prior to data acquisition. De-identified data will be posted to OSF following publication.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be made available following publication.
Access Criteria: IPD will be available on OSF to all who are interested.